CLINICAL TRIAL: NCT05020158
Title: The Family Talk Intervention in Clinical Practice When a Parent With Dependent Children or a Child is Severely Ill: An Effectiveness-implementation Study
Brief Title: The Family Talk Intervention When a Parent With Dependent Children or a Child is Severely Ill
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ersta Sköndal University College (Other)
Responsible Party: Principal Investigator, Malin Lövgren, Associate professor, Ersta Sköndal University College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Marie Cederschiöld
Record Dates: First submitted 2021-05-11; First posted 2021-08-25 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Illness Terminal
Keywords: Pediatric palliative care; Adult palliative care; Family Intervention

STUDY DESIGN:
Intervention Model Description: Pre-post effectiveness-implementation hybrid design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Family Talk intervention (Experimental): FTI entails six meetings, with intervals of 1-2 weeks between meetings. Meetings 1-2 include only the parent(s) and focus on their experiences of the situation, as well as the consequences of the diagnosis for each family member. The parent(s) will formulate the goal of the intervention. Meeting 3: Interviews will be held with each child and includes the child's life situation. Meeting 4 includes the parent(s) and focuses on planning the family meeting. The children's thoughts and questions serve as a guide for the upcoming family meeting. Meeting 5 is a family meeting and consists of questions and issues raised earlier by the family members. Meeting 6 is a follow-up with all family members. The meeting is guided by the family members' needs, e.g., regarding communication and parenting. If the intervention is interrupted unexpectedly and cannot be finished as scheduled due to extraordinary circumstances, extra meetings are available (Meetings 7-11).
  Interventions: Other: Family Talk Intervention

INTERVENTIONS:
Other: Family Talk Intervention — A psychosocial family-based intervention that is designed to give support to an entire family when a child has life-threatening illness.

SUMMARY:
The overall aim of this study is to evaluate the effects and the implementation process of the Family Talk Intervention (FTI) in clinical practice when a child or a parent of dependent children has a life-threatening/life-limiting illness (cancer, neurological diseases, etc.). During 2021, FTI will be implemented in several different care contexts including a children's hospital and a university hospital in Sweden. Social workers will be educated in using the FTI in their clinical work. This study has a pre-post effectiveness-implementation hybrid design using mixed method. Data collection will be made using web-based questionnaires and interviews with families and social workers, and observations will be performed throughout the study.

DETAILED DESCRIPTION:
The Family Talk Intervention (FTI), also called Beardslee's Family Intervention is a manual-based complex intervention and involves families who have children aged 6-18 years. The core elements are to support the families in talking about illness-related subjects, support the parents in understanding the needs of their children and how to support them, and support the families in identifying their strengths and how best to use them.

The overall aim of this trial is to evaluate the effects and the implementation process of FTI in clinical practice when a parent or a child has a life-threatening/life-limiting illness (cancer, neurological diseases, etc.). More specifically, to examine the effects of FTI regarding family communication and psychosocial health among family members (Aim 1) and describe facilitating factors and barriers for implementing FTI in everyday clinical practice (Aim 2).

The FTI has previously been pilot-tested in the context of specialized palliative home care with promising results. In pilot-tests, an assigned interventionist was used for intervention delivery, while in this continued trial, social workers will deliver the intervention as a part of their clinical work.

This trial has a pre-post effectiveness-implementation hybrid design using mixed method. It will be placed at a children's hospital and at a university hospital in Sweden and conducted by all social workers working there (n=25). Education of social workers in working with FTI will take place during 2021 and families will be invited to the project from April 2022 and until power has been reached. Data will be collected using web-based questionnaires and interviews with families and social workers, and observations will be performed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Families that include a child with a life-threatening/life-limiting illness.
* 2-3 months should have passed since diagnosis or relapse.
* <2 members of the family need to participate

Exclusion Criteria:

-

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Changed family communication from Family Adaptability and Cohesion Scale IV (FACES IV) | At baseline (before FTI starts), after the end of FTI/three months later (follow-up 1), and six months after that (follow-up 2).
  Measures family communication

SECONDARY OUTCOMES:
Changed resilience for adults measured by the Resilience Scale (RS-14) | At baseline (before FTI starts), after the end of FTI/three months later (follow-up 1), and six months after that (follow-up 2).
  Measures psychosocial health for parents/guardians and for children aged 13 years and older
Changed resilience in children measured by the Resilience Scale for Children (RS-10), | At baseline (before FTI starts), after the end of FTI/three months later (follow-up 1), and six months after that (follow-up 2).
  Measures psychosocial health for children aged 8-12 years
Changed symptoms of pathologic grief measured by Prolonged Grief Disorder (PG-12) | At baseline (before FTI starts), after the end of FTI/three months later (follow-up 1), and six months after that (follow-up 2).
  Measures pre-death grief
Generalized Anxiety Disorder (GAD) | At baseline (before FTI starts), after the end of FTI/three months later (follow-up 1), and six months after that (follow-up 2).
  Measures anxiety in adults
Changed feelings of strength and weaknesses in children measured by The Strengths and Difficulties Questionnaire (SDQ) | At baseline (before FTI starts), after the end of FTI/three months later (follow-up 1), and six months after that (follow-up 2).
  Measures self-perceived strength and weakness. Parent Proxy for children under 11 years.
Changed feelings of parental skill measured by the Parental Skill Questionnaire (SDQ) | At baseline (before FTI starts), after the end of FTI/three months later (follow-up 1), and six months after that (follow-up 2).
  Measures self-perceived parental skill
Changed key mechanisms to promote and inhibit implementation measured by The Swedish Normalization Process Theory Measure (S-NoMAD) | At baseline (after FTI education), four months later (follow-up 1) and 12 months later (follow-up 2).
  Characterizes and explains key mechanisms that promote and inhibit the implementation, embedding and integration of new health techniques, technologies and other complex interventions.
Changed organizational context measured by Alberta Context Tool (ACT) | At baseline (after FTI education), four months later (follow-up 1) and 12 months later (follow-up 2).
  Measures organizational context for use in complex healthcare settings.

CONTACTS AND LOCATIONS:
Overall Officials: Malin Lövgren, PhD, Principal Investigator — Ersta Sköndal Bräcke University College
Locations (1):
- Marie Cederschiöld University College, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thermaenius I, Holm M, Arestedt K, Udo C, Alvariza A, Lundberg T, Wallin L, Lovgren M. Implementing the Family Talk Intervention among families with a severely ill parent or child with palliative care needs- a longitudinal study of the perspectives of hospital social workers. Front Health Serv. 2025 Jun 13;5:1527431. doi: 10.3389/frhs.2025.1527431. eCollection 2025. PMID 40584244